CLINICAL TRIAL: NCT04111783
Title: Preoperative Rapid Pou Ultrasound（Pre-operative Ultrasound Evaluation Protocol） Assessment of Randomized Controlled Clinical Trials for Optimal Management of Anesthesia in Critically Ill Patients Undergoing Emergency Surgery.
Brief Title: Preoperative Rapid Pou Ultrasound Assessment in Critically Ill Patients Undergoing Emergency Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: daizhongliang-03
Record Dates: First submitted 2019-09-25; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Emergency Surgery
Keywords: anesthesia; Preoperative rapid POU ultrasound; clinical trials

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Volunteers and data collectors was masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POU ultrasound intervention test group (Experimental): The experimental group used POU protocol ultrasound to perform a heart scan and a standard scan, a large vascular scan under the xiphoid, a body cavity scan, a standard section, and a lung scan in 10 minutes. Comprehensive preoperative circulation and assessment of systemic conditions, and guided intraoperative anesthesia management with assessment results.
  Interventions: Device: POU protocol ultrasound
- Control group (No Intervention): the anesthesiologist performed according to the existing preoperative evaluation program and existing experience, and guided the anesthesia management with the evaluation results.

INTERVENTIONS:
Device: POU protocol ultrasound — The evaluation method performed a preoperative examination of the patient within 10 minutes by a heart scan and a standard scan of the face, a large vascular scan under the xiphoid, a body cavity scan, and a standard scan of the face and a lung scan. Preparation, providing anesthesia and surgeons with a fast, comprehensive and accurate preoperative judgment with important clinical and social significance.
  Arms: POU ultrasound intervention test group

SUMMARY:
With the development of society, the number of emergency critical operations is increasing year by year. Traditionally, the patient's systemic and circulatory status is indirectly assessed by testing and blood pressure heart rate. There are cases where the diagnosis is imperfect and the results are unreliable. Preoperative POU rapid ultrasound is a preoperative bedside ultrasound evaluation method first proposed by the Anesthesiology Department of Huaxi Hospital (three engineering units). This project will cooperate with Huaxi Hospital to explore whether the effect of intraoperative anesthesia management under POU guidance is better than traditional anesthesia management. This study will provide a new preoperative evaluation anesthesia management program for emergency critically ill patients with important clinical and social significance.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria, the patients will be randomly divided into two groups：In the control group, the anesthesiologist performed according to the existing preoperative evaluation program and existing experience, and guided the anesthesia management with the evaluation results.The experimental group used POU protocol ultrasound to perform a heart scan and a standard scan, a large vascular scan under the xiphoid, a body cavity scan, a standard section, and a lung scan in 10 minutes. Comprehensive preoperative circulation and assessment of systemic conditions, and guided intraoperative anesthesia management with assessment results.

ELIGIBILITY:
Inclusion Criteria:

* 1.pulse oxygen saturation (spO2) ≤ 92% when inhaling air.
* 2.respiratory frequency ≥ 20 beats / min.
* 3.systolic blood pressure (sbp) <90mmHg.
* 4.heart rate (hr)>100 times/min.
* 5.requires positive inotropic drugs and/or vasopressors.
* 6.need artificial ventilation.
* 7.Signing informed consent.

Exclusion Criteria:

* 1.age <14 years old.
* 2.unable to perform ultrasound evaluation (bandage, clam shell).
* 3.participated in other clinical trials in the first 3 months of the study.
* 4.researchers believe that it is not appropriate to include this tester.
* 5.any reason can not cooperate with this study.
* 6.cardiac surgery patient
* 7.organ transplant patient.
* 8.obstetric surgery patient.
* 9.you can start rescue after entering the room (such as CPR, etc.), and you are not allowed to perform ultrasound scans.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-29 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Severe complication rate | The follow-up period ranges from the first patient recruited to the last patient within 6 months after admission, up to 2 years
  Serious complications include cardiac arrest, respiratory failure, hemorrhagic shock, pulmonary embolism, etc.
mortality rate | The follow-up period ranges from the first patient recruited to the last patient within 6 months after admission, up to 2 years
  The number of patients who died from any cause since the date of randomization.
Subjects' health status scores 30 days, 90 days, half a year, and one year after surgery. | The follow-up period ranges from the first patient recruited to the last patient within 6 months after admission, up to 2 years
  Follow-up was performed 30 days, 90 days, half a year, and one year after surgery, and the patient's prognosis was assessed using a health score sheet.

CONTACTS AND LOCATIONS:
Overall Officials: ping wang, MD, Principal Investigator — China, Guangdong ,Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No